CLINICAL TRIAL: NCT01951963
Title: Sub-dissociative Ketamine for the Management of Acute Pediatric Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A12-158
Record Dates: First submitted 2013-09-24; First posted 2013-09-27 (Estimated); Results first posted 2017-10-16 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Pain
Keywords: pain management; ketamine; morphine; pediatrics; emergency medicine
MeSH Terms: conditions — Pain; Agnosia | interventions — Ketamine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine (Experimental): Ketamine, single dose, 0.3 mg/kg, IV
  Interventions: Drug: Ketamine
- Morphine (Active Comparator): Morphine, single dose, 0.05 mg/kg, IV
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Ketamine
  Arms: Ketamine
Drug: Morphine
  Arms: Morphine

SUMMARY:
The proposed trial is a prospective, double blinded, randomized control trial with the primary aim of determining whether a single, sub-dissociative dose of ketamine will decrease the total narcotic requirements of pediatric patients requiring intravenous analgesia in an urban emergency department (ED) compared to a group of patients who receive morphine alone for pain management. Patients are randomized to receive either a single bolus of ketamine (0.3 mg/kg) or a single bolus of morphine (0.05mg/kg). All subsequent pain management will be accomplished using morphine. Patient, family member, and research staff pain scores will be recorded, until 3 hours post study medication administration. Family members are contacted via telephone 24 hours post-ED discharge, and again at 7 days post-hospital discharge, for evaluation via Post Hospitalization Behavior Questionnaire. Narcotic equivalents will be calculated for up to 3 hours post study medication administration and compared between the ketamine and morphine groups.

ELIGIBILITY:
Inclusion Criteria:

* Age: 3-17 years old
* Condition (medical or trauma) requiring opioid pain management per standard of care
* Need to establish an IV per standard of care
* Treating physician agrees to manage the patient's pain with morphine following randomization.

Exclusion Criteria:

* Trauma Team Activation
* Known allergy to ketamine
* Family member unable/unavailable to provide informed consent
* When appropriate, patient unwilling to provide assent
* High suspicion of injury related to child abuse
* Patient and/or family member is non-English speaking
* Patient is incarcerated

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 77 (Actual)
Dates: Start 2012-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron M Burnett, MD, Principal Investigator — Regions Hospital
Locations (1):
- Regions Hospital, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
We do not have a plan to share IPD

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 77 met eligibility criteria and 63 were randomized to one of the two study groups.
Groups:
- Ketamine: Ketamine, single dose, 0.3 mg/kg, IV
  The final sample included 40 subjects, 20 in the Ketamine group. The baseline characteristics were similar between the two groups. These patients were randomized to receive a single bolus of ketamine (0.3 mg/kg). These are standard recommended pediatric weight-based analgesic doses of Ketamine. Patient weight was obtained by the treating RN using a scale or Broselow tape. A blinded 10mL syringe containing study drug was prepared and delivered to the bedside by a pharmacist. After administration of study drug all future analgesic doses were restricted to morphine and were given at the discretion of the treatment team.
- Morphine: Morphine, single dose, 0.05 mg/kg, IV
  The final sample included 40 subjects, 20 in the Morphine group. The baseline characteristics were similar between the two groups. These patients were randomized to receive a single bolus of morphine (0.05mg/kg). These are standard recommended pediatric weight-based analgesic doses of Morphine. Patient weight was obtained by the treating RN using a scale or Broselow tape. A blinded 10mL syringe containing study drug was prepared and delivered to the bedside by a pharmacist. After administration of study drug all future analgesic doses were restricted to morphine and were given at the discretion of the treatment team.
Period: Overall Study
Arm/Group | Ketamine | Morphine
Started | 31 | 32
Completed | 31 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ketamine: Ketamine, single dose, 0.3 mg/kg, IV
  The final sample included 40 subjects, 20 in the Ketamine group. Inclusion criteria was defined as, patients age 3-17 years old, medical or traumatic condition requiring intravenous opioid analgesics, ability to obtain consent from parents and assent from the patient. The baseline characteristics were similar between the two groups. These patients were randomized to receive a single bolus of ketamine (0.3 mg/kg). These are standard recommended pediatric weight-based analgesic doses of Ketamine. Patient weight was obtained by the treating RN using a scale or Broselow tape. A blinded 10mL syringe containing study drug was prepared and delivered to the bedside by a pharmacist. After administration of study drug all future analgesic doses were restricted to morphine and were given at the discretion of the treatment team.
- Total: Total of all reporting groups
Arm/Group | Ketamine | Morphine | Total
Number analyzed (Participants) | 31 | 32 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 31 | 32 | 63
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.3 (3.6) | 12.7 (3.7) | 13.0 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 19 | 23 | 42
Region of Enrollment [Number; unit: participants]
  United States | 31 | 32 | 63

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Narcotic Consumption
Description: All opioids administered were converted to morphine equivalents in milligrams (eq. mg) via standard equianalgesic calculations. Pre-study drug opioids information was also collected.The number of subjects who received a morphine dose after administration of the study drug, both within one hour or at all was included in the outcome measure results.
Time Frame: 3 hours post study drug administration
Population: The number of subjects in each group who received at least one dose of opioids post study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Ketamine: Ketamine, single dose, 0.3 mg/kg, IV
  Ketamine
  prospective, double blind, randomized control trial. After informed consent, patients 3-17 years old requiring intravenous analgesics were randomized to receive either a single dose of 0.3mg/kg ketamine or 0.05mg/kg morphine in addition to standard opioid based analgesia. These weight-based doses of Ketamine and Morphine are the standard recommended doses from the Lexicomp Drug Reference Handbook, Pediatric and Neonatal Dosing (2011-2012).
- Morphine: Morphine, single dose, 0.05 mg/kg, IV
  Morphine
  prospective, double blind, randomized control trial. After informed consent, patients 3-17 years old requiring intravenous analgesics were randomized to receive either a single dose of 0.3mg/kg ketamine or 0.05mg/kg morphine in addition to standard opioid based analgesia. These weight-based doses of Ketamine and Morphine are the standard recommended doses from the Lexicomp Drug Reference Handbook, Pediatric and Neonatal Dosing (2011-2012).
Arm/Group | Ketamine | Morphine
Number analyzed (Participants) | 31 | 32
Participants | 19 | 14

2. Primary Outcome: Adverse Drug Reaction
Description: Rate of pain medication related adverse events during their ED stay and at 24 hours post discharge from the ED. the research team will complete the Adverse Event case report form to determine any adverse events occurring during the study period. Family members will be contacted via telephone 24 hours (±8 hours) following their visit in the Emergency Department to complete the Discharge Adverse Event case report form.
Time Frame: 3 hours post study drug administration
Population: Rate of pain medication related adverse events during their ED stay and at 24 hours post discharge from the ED will be compared using unadjusted Fisher's exact of a composite measure (≤ 1 events vs. > 1).
Measure: Count of Participants; unit: Participants
Groups:
- Ketamine: Ketamine, single dose, 0.3 mg/kg, IV
  Ketamine
- Morphine: Morphine, single dose, 0.05 mg/kg, IV
  Morphine
Arm/Group | Ketamine | Morphine
Number analyzed (Participants) | 31 | 32
Participants | 2 | 3

3. Other Pre Specified Outcome: Pain Scale Rating Agreement Among Patient, Parent, and Research Staff
Description: FLACC scores were assessed on the patient using the FLACC scale (0-10) by the parent, treating RN/trained research assistant.
  * FLACC - Parents 30 Minutes Post dose
  * FLACC - Staff 30 Minutes Post dose
  Wong-Baker Faces scale is a self-assessment of pain Scale of 1-10 pain.
Time Frame: Up to 3 hours post pain medication administration
Population: Wong-Baker Faces scale is a self-assessment of pain Scale. FLACC Score (FLACC = Face, Legs, Activity, Crying and Consolability) is a behavioral observational pain rating scale that looks for specific behaviors and scores them. Both scales are scored 0-10 with 0 representing no pain. Lower scores are better outcomes.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ketamine | Morphine
Number analyzed (Participants) | 31 | 32
Scores on a scale
  FLACC - Staff 30 Minutes Post dose | 1.1 (1.7) | 1.1 (1.6)
  FLACC - Parents 30 Minutes Post dose | 2.0 (2.1) | 1.9 (1.9)
  Wong-Baker Faces pain scale changes | -3.5 (2.4) | -3.7 (2.4)

ADVERSE EVENTS:
Arm/Group | Ketamine | Morphine
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/32
Other Adverse Events (participants affected / at risk) | 2/31 | 2/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=31) | Morphine (N=32)
Allergic Reaction to study drug (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) — Rash
vomiting/nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes